CLINICAL TRIAL: NCT03550729
Title: Effects of Physical Training on Vascular Function as a Therapeutic Target in Pulmonary Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Isabel Blanco, Senior specialist in Pneumology, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TrainHAP
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Exercise training; Biomarkers
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Endurance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): 12-weeks of supervised endurance training program.
  Interventions: Behavioral: Endurance training

INTERVENTIONS:
Behavioral: Endurance training — Endurance training 3 times per week during 3 months using interval training above 70% of load peak reached in the incremental exercise test. The duration of the sessions will be adapted individually to each patient (approximately 60 minutes).

SUMMARY:
The role of physical training in the treatment of pulmonary arterial hypertension (PAH) is controversial. The aim of the project is to evaluate the effect of physical training on markers of endothelial function and integrity and to identify those biomarkers associated with a better therapeutic response in patients with PAH and in an experimental model of pulmonary hypertension. Methodology: 1) Study in humans: sample size will be 50 patients with PAH. Responders and non-responders will be identified for a 12-week resistance training program. Before and after the physical training program, endothelial microparticles and circulating vascular progenitor cells, and metabolomic and mitochondrial function parameters in circulating endothelial cells will be analyzed. Patients will be identified in whom a more favorable response to the training program is obtained. Additionally, investigators will evaluate the relationship between this response and the biomarkers both at baseline and their change with the training program. 2) Study in a murine experimental model: investigators will study mice with pulmonary hypertension induced by the administration of Semaxanib (SU5416) and exposure to hypoxia for 3 weeks and control mice. Half of them will exercise on a treadmill for 3 weeks. At the end of the program the right ventricular pressure will be measured and the animals will be sacrificed. Morphometric studies in pulmonary and cardiac tissue, pulmonary endothelial function and metabolomic parameters in cardiac and skeletal muscle will be performed. Differences in these variables between the different experimental groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Functional class of New York Heart Association (NYHA) II-III
* Diagnosis of pulmonary hypertension (PH) by right heart catheterization, as follows:
* Mean pulmonary arterial pressure (mPAP) >=25 mmHg
* Pulmonary vascular resistance (PVR) ≥240 din / s / cm5
* Pulmonary interlock pressure (PCWP) ≤15 mmHg
* Patients with optimized PAH treatment, including intensified treatment with diuretics and who have remained stable for at least 2 months before entering the study (changes in medical treatment are not expected during the entire 12-week study period)
* Be able to understand and be willing to sign the informed consent form

Exclusion Criteria:

* Other type of PH (groups 2, 3, 4 or 5)
* Pregnant women
* Disability to exercise on a cycle ergometer or walk
* Acute infection or fever
* Any change in the treatment of the disease in the last 2 months
* Acute ischemic heart disease, unstable angina pectoris, exercise-induced ventricular arrhythmias, decompensated heart failure
* History or suspicion of inability to cooperate adequately in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Endurance time | Baseline - 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Spain